CLINICAL TRIAL: NCT07021144
Title: VA|PREVENTION: Randomized Controlled Trial of a Person-Centred Digital Intervention to Prevent Diabetes in High-Risk Adults
Acronym: VA|PREVENTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Universidade Nova de Lisboa (Other); FCiências.ID - Associação para a Investigação e Desenvolvimento de Ciências (Lisbon, Portugal) (Unknown); Nursing School of Lisbon (Other); Faculdade de Motricidade Humana de Lisboa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VA|PREVENTION_01
Record Dates: First submitted 2025-05-27; First posted 2025-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pre-diabetes; Pre-diabetic State
Keywords: Diabetes Prevention via a Virtual Human Coach; Digital behaviour change intervention; Hybrid Effectiveness-Implementation Randomised Controlled Trial; Cost-Effectiveness; Type 2 Diabetes Prevention
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA|PREVENTION web app (Experimental): Participants will use the VA|PREVENTION web application as a digital health intervention, for 10 months. They will access the app via personal devices (smartphone, tablet, or computer) and use a pedometer to self-monitor physical activity by counting steps.
  Interventions: Behavioral: VA|PREVENTION web application (digital intervention)
- T2D Guidebook (Active Comparator): Participants will have access to the "Prevenção da Diabetes Tipo 2" guidebook, which provides information on diet and physical activity, along with a pedometer to self-monitor physical activity by counting steps.
  Interventions: Behavioral: Type 2 Diabetes Guidebook

INTERVENTIONS:
Behavioral: VA|PREVENTION web application (digital intervention) — VA|PREVENTION web app, a digital intervention incorporating behaviour change techniques delivered by a Virtual Human Coach (VHC), educational content and progress tracking via a dashboard.
  Arms: VA|PREVENTION web app
Behavioral: Type 2 Diabetes Guidebook — T2D prevention guidebook, an educational material that include standard guidelines on healthy eating and the importance of regular physical activity and reduction of sedentary behaviour.
  Arms: T2D Guidebook

SUMMARY:
The goal of this clinical trial is to help prevent the development of type 2 diabetes (T2D) in adults who are at risk. The study will test a digital intervention called VA|PREVENTION, a web application designed to support and promote healthy behaviour changes known has T2D risk factors, such as physical activity, diet, and sedentary behaviuor. The main questions this study will explore are:• Is the VA|PREVENTION web app, which includes a virtual human coach, effective in preventing type 2 diabetes?• Can the VA|PREVENTION web app be successfully implemented in real-world settings?• Is the VA|PREVENTION web app cost-effective?• Is it safe for participants to use?To answer these questions, the study team will compare the VA|PREVENTION web app to an openly available guidebook that provides standard information about preventing type 2 diabetes.Participants will complete the following activities:

* Participants will be randomly assigned to one of two groups: one group will use the VA|PREVENTION app, while the other group will have access to an openly accessible guidebook on T2D prevention.
* Participants will be in the study for 10 months.
* Participants will be assessed at the start of the study (baseline), and again at 4 months and 10 months.
* Assessments will include body measurements (such as weight, height, and waist circumference), physical activity levels, and responses to questionnaires.

DETAILED DESCRIPTION:
T2D risk adults will be invited by nurses and community pharmacists, leveraging their trusted roles within the healthcare system. Recruitment activities will prioritize fair treatment and respect for informed consent. Only participants fully capable of understanding the informed consent terms will be included in the study. Potential participants will receive detailed information about the study's purpose, procedures, potential risks, and benefits. After providing time for questions and discussion, written informed consent will be obtained. Following consent, participants will undergo screening to confirm eligibility according to predefined inclusion and exclusion criteria. Those meeting all eligibility criteria will proceed to the baseline visit (T0), during which initial assessments will be conducted. After the baseline assessment, participants will be randomized into one of the study groups. Following randomization, the assigned intervention will be initiated, with subsequent visits scheduled at 4 months (T1) and 10 months (T2) for data collection.Upon obtaining informed consent, participants will undergo screening to verify eligibility according to predefined inclusion and exclusion criteria. Those who meet all criteria will proceed to the baseline visit (T0), where initial assessments will be conducted. Following this, participants will be randomly assigned to one of the study groups. The assigned intervention will then be initiated, with subsequent visits scheduled at 4 months (T1) and 10 months (T2) for data collection. At these timepoints, waist circumference, the primary endpoint, as well as data on anthropometric measurements (heigh and weight), diabetes risk (FINDRISC score), dietary adherence (through MEDAS questionnaire), physical activity (through accelerometry measurements), and health resources utilization will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* FINDRISC Score ≥12 (moderate, high or very high) and/or prediabetes, defined as either:

  * HbA1c between 5.7%-6.4% within the last two years; or
  * Impaired Glucose Tolerance (IGT) based on an Oral Glucose Tolerance Test (OGTT) at the 120-minute mark, with values between 140 and 199 mg/dL in the past three years;
* Able to understand, speak and write Portuguese;
* Able to provide written informed consent;
* Access to a smartphone, tablet or computer with internet connection;
* Plan to reside in the recruitment/study area for the next 10 months

Exclusion Criteria:

* Established Type 1 and 2 Diabetes Mellitus diagnosis;
* Pregnancy - Self-reported as currently pregnant, planning to become pregnant, or not practicing contraception, in the following 10 months (if applicable);
* Conditions precluding technology use (e.g. cognitive decline, dependent upon a carer for daily activities);
* Use of anti-obesity or diabetes medication, such as Metformin, Glucagon-like peptide-1 analogue (GLP-1), or other medications known to significantly impact weight (either gain or loss), currently or within the preceding 3 months;
* Following a prescribed medical diet;
* Having undergone bariatric surgery within the past 3 years or planning surgery within the next 10 months;
* Any mental health condition, including, but not limited to, eating disorders or alcohol/substance abuse, that would impact fully participating on the study;
* Participating in a concurrent weight management program and/or relevant interventional research protocol;
* Contraindication to physical activity or weight loss;
* Existing thyroid disorder;
* Active cancer or less than 6 months from treatment;
* Unable to provide informed consent or absence of a legal representative that can provided it on behalf of the patient;
* Institutionalised adults;
* Foreseeable difficulty in attending study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in waist circumference (WC) | Baseline (T0), 4 months (T1), 10 months (T2)
  The measurement of WC will be conducted using a standardized procedure (NIH, 1994; Pimenta et al., 2015; Ross et al., 2020) with an inelastic metallic anthropometric tape. The measurement of WC will be repeated 2 times, and if the second differed more than 1 cm from the first measurement, a third measurement will be carried out. We always considered the result obtained in the second measurement unless a third measurement is carried out. If a third measurement is taken, we will consider the mode or, if mode was absent, the median value of all 3 measurements.

SECONDARY OUTCOMES:
Change in FINDRISC Score categories | Baseline (T0), 4 months (T1), 10 months (T2).
  FINDRISC risk score, is a validated tool for identifying individuals at high risk of developing T2DM. It incorporates various risk factors, including age, BMI, WC, and lifestyle habits (Lindström & Tuomilehto, 2003). Evaluating changes in FINDRISC categories allows for the assessment of the intervention's impact on overall diabetes risk, offering a comprehensive view of risk factor modification (WHO, 2020). FINDRISC risk score categories allow a maximum score of 26 points and classifies individuals into risk levels: low (< 7 points); mildly moderate (between 7 and 11 points); moderate (12-14 points); high (15-20 points) and very high (more than 20 points) (Dantas, 2017; Lindström & Tuomilehto, 2003).
Change in Body Weight and Body Mass Index | Baseline (T0), 4 months (T1), 10 months (T2)
  Body weight will be measured using a digital scale that is pre-calibrated and placed on a flat, firm surface, with participants barefoot and wearing only light clothing without accessories. Body height will be measured as the highest point of the cranium (vertex) and the horizontal surface where the individual's feet are standing, in an upright position, using a stadiometer, following a standard protocol (Gordon, Chumlea and Roche, 1988). Body mass index will be calculated using body weight (in kilograms) divided by body height squared (in meters). The measurement of body weight and height will be repeated 2 times, and if the second differed more then 0.5 kg (for weight) or 1.0 cm (for height) from the first measurement, a third measurement will be carried out. We always considered the result obtained in the second measurement unless a third measurement is carried out. When a third measurement is taken, we will consider the mode or, if mode was absent, the median value of all 3.
Change in Physical Activity and Sedentary Behaviour | Baseline (T0), 4 months (T1), 10 months (T2)
  Change in dietary behaviours will be assessed through MEDAS questionnaire. This questionnaire includes 14 items that evaluate the intake of key components of the Mediterranean diet. This is a validated tool widely used in research to assess adherence to the Mediterranean diet, which is strongly associated with reduced risk of type 2 diabetes (Martínez-González et al., 2012).
Change in Dietary Behaviours | Baseline (T0), 4 months (T1), 10 months (T2)
  Change in dietary behaviours will be assessed through MEDAS questionnaire. This questionnaire includes 14 items that evaluate the intake of key components of the Mediterranean diet. This is a validated tool widely used in research to assess adherence to the Mediterranean diet, which is strongly associated with reduced risk of type 2 diabetes (Martínez-González et al., 2012).
Quality of Life (QoL) | Baseline (T0), 4 months (T1), 10 months (T2)
  Health-related quality of life will be assessed using the EQ-5D-5L questionnaire. This instrument evaluates five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L is widely accepted in clinical research and is considered a reliable measure of health outcomes over time (Herdman et al., 2011).
Digital intervention Usage and Engagement (Adoption) | Over the course of each participant's study period (expected to be for 10 months)
  Adoption will be assessed via rates and retention, based on data collected by user and second users' interactions with the VA|PREVENTION web app. This includes:
  1. Number of complete interactions with Ema for physical activity and dietary behaviours over the intervention period;
  2. Number of complete topics answered in the educational menus;
  3. Number of visits to the dashboard: (i) educative menus usage data ; (ii) self-monitoring and goal progress features; and (iii) feature showing the number of interactions with Ema;
  4. Length of use of: i) interactions with Ema; ii) Educative Menus; and iii) Dashboard for physical activity and dietary behaviours;
  5. Frequency of use of: i) interactions with Ema; ii) Educative Menus; and iii) Dashboard for physical activity and dietary behaviours
  6. Number of secondary users that access the dashboard
  7. Number of visits of secondary users to the dashboard;
Acceptability, Appropriateness, and Feasibility of Intervention | Acceptability, Appropriateness and Feasibility questionnaire responded by users, will be assessed at the end of the study visit (T3, 10 month). Interviews will be conducted after study visits completed.
  The acceptability, appropriateness, and feasibility of the VA|PREVENTION web app will be assessed through the evaluation of:
  1. Acceptability, Appropriateness and Feasibility questionnaire responded by participants/users, secondary users and managers; Each section of the questionnaire has 4 items, responded on a 5-point likert scale, ranging from completely disagree to completely agree.
  2. Qualitative data from interviews with primary and secondary users.
  3. Qualitative date from interviews with managers of Primary Care Units and Community pharmacies; These will be telephone interviews, and thematic saturation will be used to determine the size of the samples with a minimum of 20 interviews planned for primary users, and a minimum of 10 participants for each of the remaining samples is envisaged.
Cost-effectiveness | Baseline (T0), 4 months (T1), 10 months (T2)
  Cost-effectiveness of the web app will be assessed through Incremental Cost-Effectiveness Ratio (ICER). ICER represent the ratio of the difference in costs and the difference in health outcomes. ICERs will be calculated for the comparison of the web app intervention with control group.
  The primary ICER will be computed as cost per QALY derived using utility values calculated from the EQ-5D-5L instrument. In addition, ICERs can also be reported for the relation with other secondary outcomes, such as cost per cm reduction in waist circumference, or cost per point reduction in FINDRISC risk score.
  The cost-effectiveness analysis will adopt a healthcare payer perspective.

OTHER OUTCOMES:
Rate of Adverse Events and Software Issues | Continuously, with formal assessments at 4 months (T1), 10 months (T2)
  The assessment of adverse events and software issues will focus on the identification and reporting of both serious and non-serious adverse events, as well as any deficiencies related to the investigational digital intervention. Continuous monitoring of adverse events is crucial to safeguard participant safety and maintain the integrity of the study's outcomes.

CONTACTS AND LOCATIONS:
Locations (16):
- Portugal (16):
  - USF Cova da Piedade, Almada, Almada
  - USF Rosinha, Seixal, Amora
  - USF Charneca do Sol, Almada, Charneca Da Caparica
  - USF Inovar, Almada, Corroios
  - USF Saúde Laranjeiro, Almada, Fernão Ferro
  - USF Vista Tejo, Almada, Monte Da Caparica
  - Farmácia Alvide, Alcabideche
  - Farmácia da Ramalha, Almada
  - Farmácia Largo do Coreto, Almada
  - Farmácia Nuno Álvares, Almada
  - USF São João do Pragal, Almada
  - Farmácia Romeiro, Amadora
  - Farmácia Santa Marta, Barreiro
  - Farmácia Vale Fetal, Caparica
  - USF Costa do Mar, Costa da Caparica
  - Farmácia Quinta da Luz, Lisbon

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available in an aggregated form and will not be directly linked to the participants, making it impossible to associate the data with their identity. This data will be accessible on the national open-access repository promoted by the project's funder Fundação para a Ciência e Tecnologia (FCT), known as the Polen repository. Access will public for studies previously submitted and approved by an ethics committee and are deemed relevant, allowing other researchers to use it to advance scientific research and the development of new solutions in the healthcare field.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data generated by the study will be made publicly accessible within 18 to 24 months following the completion of the project studies.
Access Criteria: Access will be granted through the Polen repository, which is provided by Portugal's national science funding agency, Fundação para a Ciência e a Tecnologia, I.P. (FCT).
URL: https://repositorio.polen.fccn.pt/

REFERENCES:
- [Background] Plan and operation of the Third National Health and Nutrition Examination Survey, 1988-94. Series 1: programs and collection procedures. Vital Health Stat 1. 1994 Jul;(32):1-407. PMID 7975354
- [Background] Pimenta NM, Santa-Clara H, Melo X, Cortez-Pinto H, Silva-Nunes J, Sardinha LB. Finding the Best Waist Circumference Measurement Protocol in Patients With Nonalcoholic Fatty Liver Disease. Nutr Clin Pract. 2015 Aug;30(4):537-45. doi: 10.1177/0884533615583092. Epub 2015 Apr 23. PMID 25908607
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Altenburg TM, Wang X, van Ekris E, Andersen LB, Moller NC, Wedderkopp N, Chinapaw MJM. The consequences of using different epoch lengths on the classification of accelerometer based sedentary behaviour and physical activity. PLoS One. 2021 Jul 15;16(7):e0254721. doi: 10.1371/journal.pone.0254721. eCollection 2021. PMID 34265011
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Migueles JH, Cadenas-Sanchez C, Ekelund U, Delisle Nystrom C, Mora-Gonzalez J, Lof M, Labayen I, Ruiz JR, Ortega FB. Accelerometer Data Collection and Processing Criteria to Assess Physical Activity and Other Outcomes: A Systematic Review and Practical Considerations. Sports Med. 2017 Sep;47(9):1821-1845. doi: 10.1007/s40279-017-0716-0. PMID 28303543
- [Background] Mikkelsen MK, Berg-Beckhoff G, Frederiksen P, Horgan G, O'Driscoll R, Palmeira AL, Scott SE, Stubbs J, Heitmann BL, Larsen SC. Estimating physical activity and sedentary behaviour in a free-living environment: A comparative study between Fitbit Charge 2 and Actigraph GT3X. PLoS One. 2020 Jun 11;15(6):e0234426. doi: 10.1371/journal.pone.0234426. eCollection 2020. PMID 32525912
- [Background] Lindstrom J, Tuomilehto J. The diabetes risk score: a practical tool to predict type 2 diabetes risk. Diabetes Care. 2003 Mar;26(3):725-31. doi: 10.2337/diacare.26.3.725. PMID 12610029
- [Background] Ross R, Neeland IJ, Yamashita S, Shai I, Seidell J, Magni P, Santos RD, Arsenault B, Cuevas A, Hu FB, Griffin BA, Zambon A, Barter P, Fruchart JC, Eckel RH, Matsuzawa Y, Despres JP. Waist circumference as a vital sign in clinical practice: a Consensus Statement from the IAS and ICCR Working Group on Visceral Obesity. Nat Rev Endocrinol. 2020 Mar;16(3):177-189. doi: 10.1038/s41574-019-0310-7. Epub 2020 Feb 4. PMID 32020062